CLINICAL TRIAL: NCT04689399
Title: Sensitivity and Specificity of SARS-CoV-2 Rapid Antigen Test Compared to RT-PCR Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Testcenter Danmark, Statens Serum Institut (Unknown); Copenhagen Emergency Medical Services (Unknown)
Responsible Party: Principal Investigator, Christian von Buchwald, Professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-19
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Rapid Antigen Test; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Citizens who have booked an appointment and shows up for a COVID-19 test at a Testcenter Denmark test center in the Capital Region are offered to participate in the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standard Q COVID-19 Ag - test, produced by SD Biosensor INC. — Alle Danish citizens tested for infection with SARS-CoV-2 by swabs in the oropharynx, and subsequently analysis of the specimens by RT-PCR test at Testcenter Danmark's test centers will be included in the study. Participants will, in addition to the oropharyngeal swab they are already schedule for, be examined by a rapid antigen test.

SUMMARY:
This project aims to investigate the sensitivity and specificity of the rapid antigen test compared to RT-PCR test performed on samples from the nasopharynx and the anterior nasal cavity and the oropharynx, respectively.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the sensitivity and specificity of correct SARS-CoV-2 test results of nasopharyngeal swabs and swabs swabs from the anterior part of the nose examined by rapid antigen test (Standard Q COVID-19 Ag - test, SD Biosensor INC.) compared with swabs from the oropharynx examined by RT-PCR test among citizens who have booked an appointment for a COVID-19 test in one of Testcenter Denmark's test centers in the Capital Region.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* A booked appointment for a COVID-19 test at one of Testcenter Denmark's test centers in the Capital Region

Exclusion Criteria:

* Previously tested positive for COVID-19
* Non-fluent in Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4697 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the rapid antigen test of COVID-19 | It is expected that the required number of participants can be included during approximately one week after t

SECONDARY OUTCOMES:
Economic analyses | It is expected that the required number of participants can be included during approximately one week after t
  We plan to calculate and compare costs of the antigen tests with the RT-PCR tests. Costs are calculated using the ingredients method, in which all components relevant to consider are included in cost estimates. The cost of the tests will include the test kit, instruments needed for testing and salaries of the personnel doing the swaps. Moreover, we will model the opportunity costs of the two alternatives (antigen tests vs. RT-PCR) in terms of their implications for number of sick days, in which patients/test takes cannot resume work. We anticipate that the antigen tests will be less expensive per positive test result and that they will have lower opportunity costs due to immediate test results instead of delayed test results.
PCR analysis on nasopharyngeal swabs | It is expected that the required number of participants can be included during approximately one week after t
  For a sample of the included patients the leftover material from the rapid antigen tests will subsequently be analyzed with the use of PCR to investigate if results diverge based on the anatomic location of the swabbed area. Patients included in the last two days of the study period (30th of December and 31th of December 2020) will be selected to have this additional analysis performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Christian von Buchwald, MD, DMSc, Professor, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No